CLINICAL TRIAL: NCT02400931
Title: The Necessity of Routine Mask Ventilation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2015-0036
Record Dates: First submitted 2015-03-23; First posted 2015-03-27 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- mask ventilation (Active Comparator): Mask ventilation will be performed before the tracheal intubation.
  Interventions: Procedure: mask ventilation; Drug: Rocuronium
- no mask ventilation (Experimental): Mask ventilation will not be performed before the tracheal intubation.
  Interventions: Procedure: no mask ventilation; Drug: Rocuronium

INTERVENTIONS:
Procedure: mask ventilation — In mask ventilation group, rocuronium of 0.6 mg/kg will be administered after the loss of consciousness. Mask ventilation wil be performed until there is no response on the train-of-four stimulus. No mask ventilation - In no mask ventilation group, rocuronium of 1.2 mg/kg will be administered after the loss of consciousness. Tracheal intubation will be performed after confirmation of no response on the train-of-four stimulus. The mask ventilation will not be performed before the tracheal intubation.
  Arms: mask ventilation
Procedure: no mask ventilation
  Arms: no mask ventilation
Drug: Rocuronium

SUMMARY:
The mask ventilation is a necessary procedure to provide oxygenation before the tracheal intubation although the gastric insufflation occurs during the mask ventilation. Sugammadex, which is recently introduced, enables the use of high-dose muscle relaxant without concerning the delayed recovery of neuromuscular blockade. It seems that there is no need to perform the mask ventilation in adults with normal airway if the investigators use high-dose muscle relaxant for the anesthetic induction because adequate muscle relaxation can be achieved within 1-2 minutes. Therefore, the investigators hypothesized that routine mask ventilation is not needed in adult patients with normal airway. The investigators will compare the incidence of desaturation and gastric insufflation between the patients with mask ventilation and the patients without mask ventilation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of age over 20 years for scheduled surgery with more than one and a half hours under general anesthesia

Exclusion Criteria:

* anticipated difficult mask ventilation,
* anticipated difficult intubation,
* ASA class 3 or 4,
* preoperative saturation less than 92%.,
* saturation less than 98% after preoxygenation
* body mass index over 35 kg/m2,
* obstructive sleep apnea,
* mass in the oral cavity or in the trachea,
* pregnant woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2015-11-23 (Actual); Study Completion 2015-11-23 (Actual)

PRIMARY OUTCOMES:
Desaturation (saturation less than 95%) | until 2 minutes after the completion of tracheal intubation
  Primary outcome is the incidence of desaturation. Desaturation is defined as the saturation less than 95% which occurs after the anesthetic induction and before the first attempt of tracheal intubation.

SECONDARY OUTCOMES:
gastric insufflation (observe the antral area of the stomach using ultrasonography) | until 2 minutes after the completion of tracheal intubation
  Secondary outcome is the antral area of the stomach. We will observe the antral area of the stomach using ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea